CLINICAL TRIAL: NCT01206426
Title: Identification of Genetic Determinants of Response to Neoadjuvant Cisplatin-based Chemotherapy in Urothelial Cancer
Brief Title: Genetic Determinants of Response to Neoadjuvant Cisplatin-based Chemotherapy in Urothelial Cancer
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 09-288-B
Record Dates: First submitted 2010-09-13; First posted 2010-09-21 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Urothelial Cancer
Keywords: Urothelial, cancer, cisplatin, neoadjuvant, chemotherapy, germline
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (germline) and tumor tissue samples will be used to perform genetic analysis. The purpose of this analysis is to determine whether a set of "cisplatin susceptibility" polymorphisms predict complete pathologic response to cisplatin-based chemotherapy and to identify novel determinants which may predict response to cisplatin-based chemotherapy.
  Samples will be biobanked for future analysis of genetic determinants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is observational clinical trial to study adult urothelial cancer patients treated with cisplatin-based neoadjuvant chemotherapy.

Hypothesis: Identification of genetic and molecular "cisplatin susceptibility" biomarkers will allow identification of urothelial cancer patients most likely to benefit from cisplatin-based neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
In this trial patients will submit germline (blood) and tumor tissue samples as part of two existing sample collection protocols for analysis of genetic and molecular markers governing response to chemotherapy. Pathologic review of tissue samples after neoadjuvant therapy will allow determination of the complete response rate (pT0 rate) and this will be compared between patients with "susceptible" and "resistant" genetic/molecular cisplatin susceptibility variants.

Primary Endpoint: Analysis of whether a small set of previously-identified germline "cisplatin susceptibility" polymorphisms associate with achievement of a complete pathologic response to neoadjuvant cisplatin-based chemotherapy in urothelial cancer patients.

Secondary Endpoints: To perform companion genetic or molecular analyses of other previously-identified gene, SNP, or microRNA "cisplatin susceptibility" candidates in these patients, using tumor and/or germline tissue.

Exploratory Endpoints: To perform unbiased, hypothesis-generating SNP, gene, or microRNA array studies to identify novel germline or tumor determinants which may predict response to cisplatin-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical T2 through T4 urothelial carcinoma of the bladder or upper tract.
* Patients must be deemed appropriate by the treating physician to require cisplatin-based neoadjuvant chemotherapy for urothelial cancer. Consideration of regional nodal status as part of the decision for appropriateness for neoadjuvant chemotherapy will be left to the treating physician.
* Patients must be scheduled to proceed to definitive urothelial cancer surgery, including either cystectomy or nephrectomy/ureterectomy, after chemotherapy.
* Age >18 years.

Exclusion Criteria:

* Patients receiving cisplatin-based chemotherapy for urothelial cancer in the adjuvant setting or for metastatic disease.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients who are about to begin neoadjuvant cisplatin-based chemotherapy for urothelial cancer and who have consented to IRB approved protocols #15550B and/or TRIDOM (IRB #14104B).
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Genetic Determinants of pT0 Status | 3 years
  To perform genetic analysis of germline samples from these patients to determine whether a set of "cisplatin susceptibility" polymorphisms predict complete pathologic response to cisplatin-based chemotherapy.

SECONDARY OUTCOMES:
Molecular Determinants of pT0 Status | 3 years
  To perform companion genetic or molecular analyses of other previously-identified gene, SNP, or microRNA "cisplatin susceptibility" candidates in these patients, using tumor or germline tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H O'Donnell, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States